CLINICAL TRIAL: NCT00338585
Title: Phase 3, Multicenter, Multi-National, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Alfimeprase in Subjects With Acute Peripheral Arterial Occlusion (NAPA-3)
Brief Title: Study of Alfimeprase's Ability to Dissolve Blood Clots in the Leg and Help Prevent the Need for Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based upon preliminary safety and efficacy results from a similar study.
Sponsor: ARCA Biopharma, Inc. (Industry)
Responsible Party: Brian Kersten, PhD, Nuvelo, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA007; NAPA-3
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Arterial Occlusive Diseases
Keywords: PAO; acute peripheral arterial occlusion; thrombolysis; blood clot; leg attack; alfimeprase; thrombus; embolism; thromboembolism; claudication; thrombolytic; thrombosis; plasminogen activator; arterial flow
MeSH Terms: conditions — Arterial Occlusive Diseases; Thrombosis; Embolism; Thromboembolism; Intermittent Claudication | interventions — alfimeprase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: alfimeprase

SUMMARY:
The purpose of this study is to directly compare the safety and efficacy of intra-thrombus alfimeprase 0.3 mg/kg with placebo in acute peripheral arterial occlusion (PAO) as measured by a 30 day open vascular free surgery rate.

DETAILED DESCRIPTION:
There is an unmet medical need to improve thrombolytic therapy in acute peripheral arterial occlusion (PAO). Currently used plasminogen activators can result in increased circulating levels of plasmin that result in a systemic "lytic state" that does not distinguish between physiologic and pathologic thrombosis. In general, mean plasminogen activator infusion durations of greater than 24 hours in order to achieve successful thrombolysis are problematic in a disease where delayed restoration of arterial flow can lead to irreversible ischemic damage. A direct thrombolytic agent like alfimeprase, with a rapid mechanism of action and a potentially safer bleeding risk profile, could facilitate a rapid restoration of arterial flow and avoidance of open vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Arteriographically confirmed acute PAO of the lower extremity with onset of symptoms within 14 days prior to randomization
* Acute index limb ischemia classified as SVS/ISCVS Class I or IIa caused by occlusion of a native artery and/or bypass graft (vein or prosthetic). Only Class I subjects with abrupt onset of ischemic rest pain or abrupt onset/progression of lifestyle-limiting claudication are eligible
* Acute PAO with a need for urgent surgical intervention to restore arterial blood flow in the event of unsuccessful thrombolytic therapy
* Available for follow-up assessments

Exclusion Criteria:

* Contraindication to systemic anticoagulation
* History of endovascular procedure or open vascular surgery on the index limb within the past 30 days
* History of significant acute or chronic kidney disease that would preclude contrast angiography
* Known allergy to contrast agents
* History of heparin induced thrombocytopenia
* Participation in any study of an investigational device, medication, biologic, or other agent within 30 days prior to randomization
* Any thrombolytic therapy within 5 days prior to randomization
* Past participation in any alfimeprase trial
* Pregnant, lactating, or actively menstruating women or women of childbearing potential who are not using adequate contraceptive precautions
* Investigator inability to advance guidewire through index occlusion
* Any other subject feature that in the opinion of the investigator should preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2006-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

SECONDARY OUTCOMES:
rate of arterial flow restoration
rate of improvement in index limb ABI
change in WIQ functional status scores
AEs and SAEs
major bleeding events
ICH
peripheral arterial embolic events
all cause mortality
surgical and endovascular procedures
amputation
changes in chemistry, hematology, and coagulation parameters based on central laboratory measurements
anti-alfimeprase antibody

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hirmand, MD, Study Director — ARCA Biopharma, Inc.
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- See also: Company Website — http://www.Nuvelo.com